CLINICAL TRIAL: NCT00247507
Title: The Effects of Acetylcysteine on Alleviating Damage of Oxidative Stress in Hemodialysis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 94029
Record Dates: First submitted 2005-10-31; First posted 2005-11-02 (Estimated); Last update posted 2006-10-18 (Estimated); Status verified 2005-10

CONDITIONS: Anemia; Atherosclerosis; End-Stage Renal Disease; Oxidative Stress; Pro-Inflammation
Keywords: Anemia; atherosclerosis; End-stage renal disease; Erythropoietin; Hemodialysis; Oxidative stress; Pro-inflammation
MeSH Terms: conditions — Anemia; Atherosclerosis; Kidney Failure, Chronic | interventions — Acetylcysteine

INTERVENTIONS:
Drug: acetylcysteine

SUMMARY:
The aim of this study is to explore and identify the effects of acetylcysteine, a common mucolytic with anti-oxidant property, on alleviating the damage caused by increased oxidative stress in hemodialysis patients.

DETAILED DESCRIPTION:
Oxidative stress in patients with renal failure is higher than in healthy controls. Once undergoing hemodialysis (HD) therapy, patients with end-stage renal disease even have more oxidative stress. Reactive oxygen species (ROS) denature the vital molecules, such as lipids, proteins, and nucleic acids.

Increased ROS produce oxidized low-density lipoproteins (ox-LDL), which, in turn, induce atherosclerosis and subsequent cardiovascular disease. Cardiovascular disease is the leading cause of death of HD patients. On the other hand, ROS damage RBC membrane and cause hemolysis. Hemolysis exaggerates uremic anemia and results in resistance to erythropoietin (EPO) therapy.

Acetylcysteine, a common mucolytic, is an antioxidant as well. In vivo experiments, acetylcysteine has been demonstrated to inhibit the production of ox-LDL by ROS. Acetylcysteine has also been shown as an effective drug for prevention of contrast media-induced nephropathy in high-risk patients.

Thus we hypothesize HD patients taking acetylcysteine may have less ox-LDL produced by ROS and, consequently, lower risk of cardiovascular disease. Moreover, having less damage to RBC membrane by ROS, HD patients taking acetylcysteine may have milder anemia and better responsiveness to erythropoietin therapy. Therefore, we plan to conduct a prospective trial, in which acetylcysteine is administrated to the enrolled HD patients for three months. The primary goals of the study are to realize the changes of 1) plasma ox-LDL levels, 2) the anemia status, 3) the responsiveness to EPO therapy, and 4) severity of atherosclerosis. The secondary goals are to identify the changes of oxidative stress and pro-inflammatory status in the patients.

ELIGIBILITY:
Inclusion Criteria:

* On HD thrice a week at our HD unit for more than three months
* Informed consent
* The dose of EPO and iron supplement is stationary in the previous one month
* No taking acetylcysteine in previous one month
* No using vitamin E-bonded dialysis membrane

Exclusion Criteria:

* Severe liver disease (AST or ALT >40 IU/L), proven malignancy, and severe cardiovascular disease (proved by cardiac catheter or echography examination)
* Active infection or hospitalization in previous one month
* Clinically significant bleeding episode in previous one month
* Taking vitamin C, vitamin E or other known antioxidants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-09; Study Completion 2005-12

PRIMARY OUTCOMES:
the changes of plasma ox-LDL levels
the changes of anemia status
the responsiveness to EPO therapy and severity of atherosclerosis

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Ping Hsu, M.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Pan-Chiao, Taipei, Taiwan